CLINICAL TRIAL: NCT04386590
Title: Including Manual Therapy in Pulmonary Rehabilitation Programs for US Veterans With Moderate Chronic Obstructive Pulmonary Disease: A Feasibility Study
Brief Title: Manual Therapy in Addition to Pulmonary Rehabilitation in Moderate Chronic Obstructive Pulmonary Disease.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canandaigua VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Dougherty, DC, Staff Chiropractor, Canandaigua VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1474325
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Obstructive Pulmonary Disease Moderate
Keywords: manual therapy; respiratory therapy
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Twenty Veterans between the ages of 50 and 70 years with moderate COPD, will be randomly allocated to two equal groups. Group 1: 'sham' manual therapy plus pulmonary rehabilitation program; Group 2: Chiropractic manual therapy group plus the same pulmonary rehabilitation program (CMT+PR). Participants in both groups will undergo 8 treatment sessions over a 4 week period plus an additional assessment session at week 8. All sham manual therapy and CMT will be delivered just prior to pulmonary rehabilitation.
Who Masked: Outcomes Assessor
Masking Description: Assessor will evaluate a de-identified database with the interventions labeled as 1 and 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Sham' manual therapy plus Pulmonary Rehabilitation (PR) (Sham Comparator): Treadmill walking, upper body exercise machine, light weight training and bicycle. These exercises are supervised. In addition to the standard exercise therapy, all participants will undergo a 20-minute session consisting of discussion with the patient and 11 minutes of detuned ultrasound, which has been used in previous studies to account for time and attention for the patient. The detuned ultrasound procedure is to apply the ultrasound gel and turn the machine on, but set the intensity at zero (0) W/cm2
  Interventions: Other: Sham Intervention
- Manual therapy plus Pulmonary Rehabilitation (CMT+ (Experimental): Manual therapy is made up of gentle Effleurage and cross-fibre friction massage applied to the muscles of the posterior chest wall. Manual Therapy consists of two separate manipulations (Grade V mobilization). Each manipulation involves the delivery of a high-velocity low amplitude (HVLA) posterior to anterior force directed at the inter-vertebral, costo-vertebral and costo-transverse joints. The first manipulation is delivered at the level of the upper/middle thoracic spine while the second is at the level of the middle/lower thoracic spine. In addition to the MT, the participant will also undergo Pulmonary Rehab as previously described.
  Interventions: Other: Manual Therapy Plus Pulmonary Rehabilitation

INTERVENTIONS:
Other: Manual Therapy Plus Pulmonary Rehabilitation — Manual therapy combined with Pulmonary Rehabilitation
  Arms: Manual therapy plus Pulmonary Rehabilitation (CMT+
Other: Sham Intervention — Detuned US plus Pulmonary Rehabilitation
  Arms: 'Sham' manual therapy plus Pulmonary Rehabilitation (PR)

SUMMARY:
The aim of this study is to investigate the feasibility of administering this combination of interventions (CMT plus PR) to Veterans with moderate COPD within the context of a hospital-based outpatient pulmonary rehabilitation program.

DETAILED DESCRIPTION:
In 2016, the US Congress directed the Department of Defense to initiate a program to improve the health and well-being of all military Veterans, challenging the research and scientific communities to find original ideas that "foster new directions in research and clinical care". One of the areas identified as a priority under this initiative was 'Respiratory Health'.

Chronic obstructive pulmonary disease (COPD) is a major cause of disability, hospital admission and premature death. Current management strategies have not been successful in altering the loss of lung function typically seen as the disease progresses. Results from recent pilot trials suggest the novel combination of chiropractic manual therapy (CMT) and pulmonary rehabilitation (PR) has the potential to alter the typical pattern of decline in lung function.

The aim of this study is to investigate the feasibility of administering this combination of interventions (CMT plus PR) to Veterans with moderate COPD within the context of a hospital-based outpatient pulmonary rehabilitation program.

Twenty Veterans between the ages of 50 and 70 years with moderate COPD, will be randomly allocated to two equal groups. Group 1: 'sham' manual therapy plus pulmonary rehabilitation program; Group 2: Chiropractic manual therapy group plus the same pulmonary rehabilitation program (CMT+PR). Participants in both groups will undergo 8 treatment sessions over a 4 week period plus an additional assessment session at week 8. All sham manual therapy and CMT will be delivered just prior to pulmonary rehabilitation.

The primary purpose of the study is to assess the feasibility of conducting a larger randomized controlled trial by assessing the ability to recruit, enroll, deliver interventions and collect outcome measures on Veterans with moderate COPD. Secondary outcomes include lung function (Forced expiratory volume in the 1st second: FEV1 and Forced vital capacity: FVC), exercise capacity (six-minute walking test: 6MWT), quality of life (St Georges Respiratory Questionnaire: SGRQ), anxiety and depression levels (Hospital Anxiety and Depression scale: HAD) and frequency of exacerbations. All outcome measurements will be taken by blinded assessors.

Collecting outcome measurements at 8 weeks (4 weeks after intervention has ceased) will assess the feasibility of getting Veterans to return for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male and Female
* Age range: 50-70 years
* Disease status: Moderate COPD (FEV1% predicted: moderate 50-80% (GOLD 2018))
* Concomitant disease status: Stable COPD (no exacerbations in preceding 6 months) Non-smoking (for preceding 6 months)
* Willingness to give written informed consent.
* Willingness to participate in and comply with the study requirements.

Exclusion Criteria:

* Inability to complete 6-minute walking test unassisted
* Contra-indicated to thoracic spinal manipulation

  * Thoracic joint instability
  * Acute pain on thoracic joint range of motion testing
  * High level of anxiety related to receiving thoracic spinal manipulation
* Inability to understand English
* People with a cognitive impairment, an intellectual disability or a mental illness
* Completed a pulmonary rehabilitation program in the previous 12 months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-11-02 (Estimated)

PRIMARY OUTCOMES:
Spirometry | Change from Baseline to Post Intervention (4 weeks post baseline)
  Lung function (Forced expiratory volume in the 1st second: FEV1 and forced vital capacity: FVC) will be assessed using spirometry.

SECONDARY OUTCOMES:
6 Minute Walking Test (6MWT) | Change from baseline to post intervention (4 weeks post baseline)
  Exercise capacity will be assessed using a six-minute walking test (6MWT) where capacity is determined by the total distance walked in a period of six minutes. Greater walking distance indicates greater functional capacity.
St Georges Respiratory Questionnaire: SGRQ | Change from baseline to post intervention (4 weeks post baseline)
  Quality of life questionnaire for those with COPD. Scores are calculated for three domains: Symptoms, activity and Impacts (psychosocial) and total score. Higher scores indicate more limitations.
Hospital Anxiety and Depression scale: HAD | Change from baseline to post intervention (4 weeks post baseline)
  Questionnaire assessing anxiety and depression in outpatient hospital setting. Higher scores indicate greater levels of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Dougherty, DC, Principal Investigator — VA Finger Lakes Healthcare System
Locations (1):
- Syracuse VA Medical Center, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No
Due to the phase of this study, the data will be utilized to inform the design of a larger clinical trial. Data from the larger study will be available to share de-identified data.